CLINICAL TRIAL: NCT03238261
Title: CHEMOTHERAPY AND CONCOMITANT RADIOTHERAPY VS. RADIOTHERAPY IN THE TREATMENT OF PATIENTS WITH STAGE IIIB UTERINE CANCER
Brief Title: Chemotherapy / Radiotherapy in Uterine Cervical Neoplasms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia, Columbia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: C41030310-023
Record Dates: First submitted 2017-07-31; First posted 2017-08-03 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-07

CONDITIONS: Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy and concomitant radiotherapy (Experimental)
  Interventions: Radiation: Chemotherapy and concomitant radiotherapy
- Radiotherapy (Active Comparator)
  Interventions: Radiation: Chemotherapy and concomitant radiotherapy

INTERVENTIONS:
Radiation: Chemotherapy and concomitant radiotherapy — Radiotherapy (teletherapy + high or low rate brachytherapy)

SUMMARY:
Compare the use of radiotherapy and concomitant chemotherapy, with the single use of radiotherapy in the treatment of patients with stage IIIB uterine cancer, having as an outcome the three year survival rate, the disease free survival rate, the locoregional control of the disease and the security of the treatments provided.

Specific objectives

1. Describe and compare the demographic and clinical characteristics of both groups.
2. Compare the three year survival rate in both groups.
3. Compare the response to treatment in terms of locoregional control of the disease.
4. Compare the appearance of severe and non severe adverse events directly related to the treatment in both intervention groups.

DETAILED DESCRIPTION:
Inclusion criteria Women between 18 and 80 years old, diagnosed with uterine squamous cell cancer or stage IIIB adenocarcinoma (FIGO) with ECOG equal 1 or less and a Karnofsky equal or more than 70%.

Exclusion criteria Having a concomitant or previous neoplasia, except for patients with skin tumors not associated to melanomas, platelet count under 100.000, hemoglobin levels of 10 gr/dl or above before starting the first radiotherapy session, patients with recurrent invasive uterine carcinoma, patients with compromised para aortic lymph nodes, patients with active and non controlled pelvic infection by the beginning of the treatment, creatinine depuration less than 45 ml/min confirmed with glomerular filtration rate less than 45 ml/min, neutrophils count less than 1,500/ml, and pregnant or nursing woman.

Analysis The descriptive statistical analysis will be made with proportions for the categorical variables, and for numerical variables will be made with averages, medians, standard deviations and ranges. The comparison between categorical variables will be made with square Ji proof or exact Fisher's proof when square Ji proof doesn't meet the criteria. The comparison among continuous variables with normal distribution will be established with T student distribution proof or ANOVA, and Mann-Whitnew or Kruskall proofs will be used for variables that doesn't have this type of distribution.

For the three survival rate, the Kaplan Meier method will be applied, and the survival curves will be compared with the logarithmic range proof. The Cox proportional hazard model is going to be used for the multivariate analysis and to stablish reasons. Additionally 5 interim analysis will be made.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 80 years old, diagnosed with uterine squamous cell cancer or stage IIIB adenocarcinoma (FIGO) with ECOG equal 1 or less and a Karnofsky equal or more than 70%.

Exclusion Criteria:

* Having a concomitant or previous neoplasia, except for patients with skin tumors not associated to melanomas, platelet count under 100.000, hemoglobin levels of 10 gr/dl or above before starting the first radiotherapy session, patients with recurrent invasive uterine carcinoma, patients with compromised para aortic lymph nodes, patients with active and non controlled pelvic infection by the beginning of the treatment, creatinine depuration less than 45 ml/min confirmed with glomerular filtration rate less than 45 ml/min, neutrophils count less than 1,500/ml, and pregnant or nursing woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2012-02-01 (Actual); Study Completion 2016-05-01 (Actual)

PRIMARY OUTCOMES:
Survival rate | 3 years
  the disease free survival rate

SECONDARY OUTCOMES:
The response to treatment in terms of locoregional control of the disease | 3 years
  efficacy
Events adverse | 3 years
  4. Compare the appearance of severe and non severe adverse events directly related to the treatment in both intervention groups.

IPD SHARING:
Plan to Share IPD: No